CLINICAL TRIAL: NCT05532319
Title: Phase II Trial of Hepatic Arterial inFusion Chemotherapy Sequential transaRterial Embolization cOmbined With leNvatinib and Tislelizumab in Unresectable Hepatocellular Carcinoma (FRONT Trial)
Brief Title: HAIC Sequential TAE Combined With Lenvatinib and Tislelizumab in Unresectable HCC
Acronym: FRONT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRONT-1
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Liver Cancer
Keywords: hepatocellular carcinoma; hepatic arterial infusion chemotherapy; lenvatinib; tislelizumab
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — lenvatinib; tislelizumab

STUDY DESIGN:
Intervention Model Description: The aim of this study is to evaluate the safety and efficacy of hepatic arterial infusion chemotherapy (HAIC) sequential transarterial embolization combined with lenvatinib and tislelizumab in patients with unresectable hepatocellular carcinoma (HCC), and to explore the optimal benefit population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAIC sequential TAE combined with lenvatinib and tislelizumab (Experimental): The aim of this phase II trial is to evaluate the safety and efficacy of hepatic arterial infusion chemotherapy (HAIC) sequential transarterial embolization combined with lenvatinib and tislelizumab in patients with unresectable hepatocellular carcinoma (HCC), and to explore the optimal benefit population.
  Interventions: Combination Product: HAIC sequential TAE combined with lenvatinib and tislelizumab

INTERVENTIONS:
Combination Product: HAIC sequential TAE combined with lenvatinib and tislelizumab — Patients with unresectable hepatocellular carcinoma will receive hepatic arterial infusion chemotherapy (HAIC) sequential transarterial embolization combined with lenvatinib and tislelizumab.

SUMMARY:
Patients with unresectable hepatocellular carcinoma will receive hepatic arterial infusion chemotherapy (HAIC) sequential transarterial embolization combined with lenvatinib and tislelizumab.

DETAILED DESCRIPTION:
In recent years, more and more studies have found that the efficacy of hepatic arterial infusion chemotherapy (HAIC) alone or combined with targeted drugs (such as lenvatinib) in the treatment of advanced HCC is significantly better than that of targeted monotherapy. The principle of HAIC is that chemotherapeutic drugs are continuously pumped through the hepatic artery through a microcatheter, thereby killing tumor cells and causing tumor shrinkage and necrosis. Although continuous infusion of chemotherapeutic drugs through the hepatic artery can significantly improve the local drug concentration in the tumor, and reduce the toxic and side effects of drugs on the whole body while improving the therapeutic effect, the effect of HAIC is slow. The blood supply of HCC is 95%-99% from the hepatic artery, and abundant blood supply is conducive to the continuous growth of HCC. If transarterial embolization (TAE) can be used to block the blood supply of HCC immediately after HAIC treatment, theoretically, it should further promote the effect of HAIC on tumor cell necrosis, make the tumor quickly reach PR or even CR, obtain the opportunity of hepatic resection, and finally prolong patients' survival time. However, there is still a lack of literature reports on HAIC sequential TAE in the treatment of advanced HCC. Therefore, this project intends to carry out a prospective phase II clinical study to explore the safety and efficacy (ORR, DOR, PFS, OS) of HAIC sequential TAE combined with targeted (lenvatinib) and immunotherapy (tislelizumab) quadruplets, and to screen the best benefit population.

ELIGIBILITY:
Inclusion Criteria:

* HCC is diagnosed in accordance with the clinical diagnostic criteria of the Guidelines for the Diagnosis and Treatment of primary liver Cancer (2019 edition) issued by the Health Commission of the People's Republic of China or by histopathology;
* ECOG PS 0 or 1;
* Child-Pugh A liver function;
* Chinese Liver Cancer (CNLC) stage IIb, IIIa and IIIb patients, or CNLC stage Ib and IIA patients who cannot undergo hepatectomy for various reasons;
* Expected survival time ≥6 months;
* HCC patients with incomplete portal vein obstruction or complete portal vein obstruction with abundant compensatory collateral vessels;
* Hematological indicators should meet the following conditions: hemoglobin ≥90 g/L; absolute neutrophil count ≥1.5×10^9/L; platelets ≥80×10^9/L; total bilirubin ≤1.5×ULN; ALT 3 x ULN or less; AST 3 x ULN or less; alkaline phosphatase ≤2.5×ULN; serum albumin ≥28 g/L; serum creatinine ≤1.5×ULN;
* Urinary protein <2+ or 24 h urinary protein < 1.0 g;
* For women of reproductive age, use of contraception (e.g. intrauterine devices, tablets or condoms) is required during the course of the clinical trial until 120 days after the end of the clinical trial; Women of childbearing age had negative serum or urine HCG test results within 7 days before enrollment in the study; male patients with potential reproductive partners should use effective contraception during the study period and for 120 days after the study.

Exclusion Criteria:

* Previous or co-existing other malignancies except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
* Previously received HAIC, TACE, TAE, radiofrequency ablation and other local treatments for HCC;
* Patients who have received or are using one of the following three drugs in the previous 6 months: ① immune checkpoint inhibitors, including but not limited to artemizumab, nivolumab, pembrolizumab, camrelizumab, sintilimab, toripalimab, and tislelizumab; ② molecular targeted therapy, including but not limited to sorafenib, lenvatinib, apatinib, regorafenib, anlotinib, bevacizumab, etc. ③ systemic chemotherapy drugs (such as doxorubicin, oxaliplatin, 5-FU, S-1, etc.);
* Having a congenital or acquired immunodeficiency disease (e.g. being HIV positive);
* Active infection, or body temperature ≥ 38.5℃ or white blood cell count > 15 x 10^9/L 7 days before enrollment;
* Within 3 months of enrollment, patients with hemorrhagic diseases (including but not limited to moderate/severe esophageal and gastric variceal bleeding, gastrointestinal bleeding, hemorrhagic gastric ulcer, hemoptysis > 2.5 mL per day; For positive cases of fecal occult blood, occult blood should be reexamined, and gastroenteroscopy should be performed if necessary);
* Arterial or venous thrombosis within 6 months, such as cerebrovascular accident (transient ischemic attack, cerebral hemorrhage, cerebral infarction, etc.), deep vein thrombosis, pulmonary infarction, etc.;
* Those who have a history of alcohol or psychotropic drug abuse and are unable to abstain or have mental disorders;
* Pregnant or lactating women;
* Active autoimmune diseases or previous autoimmune diseases (such as autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, etc.);
* Being treated with immunosuppressive agents or glucocorticoids (>10mg prednisone/day) within 2 weeks;
* Complicated with hepatic encephalopathy or brain metastasis;
* Medically uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg) (based on the average of BP readings obtained from ≥2 measurements);
* Uncontrolled heart disease or symptoms (including but not limited to cardiac function grade II or above, unstable angina pectoris, myocardial infarction in the previous 1 year, supraventricular or ventricular arrhythmias requiring treatment or intervention);
* Abnormal coagulation (INR > 2.0, PT > 16 s), bleeding tendency or need for thrombolytic therapy or anticoagulant therapy (although prophylactic use of low-dose aspirin or low molecular weight heparin is permitted);
* Hereditary or acquired blood diseases (e.g. hemophilia, thrombocytopenia, coagulopathy, etc.);
* Urinary protein ≥ ++ and 24-hour urinary protein 1.0 g in urine routine;
* Patients with bone metastases requiring surgical treatment for bone metastases;
* Known hypersensitivity to active ingredients or excipients contained in the study drugs (tislelizumab, lenvatinib), or a history of severe allergy to any other monoclonal antibody or antiangiogenic targeted drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
  The primary end-point is the progression-free survival rate per RECIST at six months

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival at two years will be evaluated.
objective response rate | 6 months
  Objective response rate per RECIST will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Le-Qun Li, PhD, Study Director — Guangxi Medical University Cancer Hospital
Locations (1):
- Guangxi Medical University Cancer Hospital, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No
The data underlying this study will be shared on reasonable request to the corresponding author.

REFERENCES:
- [Background] Lai Z, He M, Bu X, Xu Y, Huang Y, Wen D, Li Q, Xu L, Zhang Y, Wei W, Chen M, Kan A, Shi M. Lenvatinib, toripalimab plus hepatic arterial infusion chemotherapy in patients with high-risk advanced hepatocellular carcinoma: A biomolecular exploratory, phase II trial. Eur J Cancer. 2022 Oct;174:68-77. doi: 10.1016/j.ejca.2022.07.005. Epub 2022 Aug 15. PMID 35981413
- [Background] Li QJ, He MK, Chen HW, Fang WQ, Zhou YM, Xu L, Wei W, Zhang YJ, Guo Y, Guo RP, Chen MS, Shi M. Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin Versus Transarterial Chemoembolization for Large Hepatocellular Carcinoma: A Randomized Phase III Trial. J Clin Oncol. 2022 Jan 10;40(2):150-160. doi: 10.1200/JCO.21.00608. Epub 2021 Oct 14. PMID 34648352
- [Background] He M, Li Q, Zou R, Shen J, Fang W, Tan G, Zhou Y, Wu X, Xu L, Wei W, Le Y, Zhou Z, Zhao M, Guo Y, Guo R, Chen M, Shi M. Sorafenib Plus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib Alone for Hepatocellular Carcinoma With Portal Vein Invasion: A Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):953-960. doi: 10.1001/jamaoncol.2019.0250. PMID 31070690
- [Background] Lyu N, Wang X, Li JB, Lai JF, Chen QF, Li SL, Deng HJ, He M, Mu LW, Zhao M. Arterial Chemotherapy of Oxaliplatin Plus Fluorouracil Versus Sorafenib in Advanced Hepatocellular Carcinoma: A Biomolecular Exploratory, Randomized, Phase III Trial (FOHAIC-1). J Clin Oncol. 2022 Feb 10;40(5):468-480. doi: 10.1200/JCO.21.01963. Epub 2021 Dec 14. PMID 34905388